CLINICAL TRIAL: NCT05665582
Title: Family Members Affected by Substance Use Disorder: How do They Cope and What Are Their Expressed Needs for Support?
Brief Title: Family Members Affected by Substance Use Disorder - a Follow-up Study
Status: Completed | Type: Observational
Sponsor: Sorlandet Hospital HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: SSHF_58-04
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2016-01

CONDITIONS: Caregiver Burden
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Affected family members of patients with Substance use disorders: The family sample was recruited from at a Norwegian addiction treatment unit where close relatives of patients in treatment for SUD participated in a family program.
  Interventions: Other: Family program

INTERVENTIONS:
Other: Family program — A 4-day psychoeducational family program.

SUMMARY:
The present study registration relates to a quantitative sub-study of a larger mixed method study, including also a qualitative sub-study. Together, these investigations will provide complementary insights. The quantitative study is a follow-up study of close relatives (> 16 years) of patients in treatment for substance use disorder (SUD) who participated in a group-based 4-day psychoeducational program.

DETAILED DESCRIPTION:
The study is a follow-up study of close relatives (> 16 years) of patients in treatment for SUDs who participated in a group-based 4-day psychoeducational program. The investigators will examine whether the family intervention in the specialized treatment services has benefits in terms of typical patient reported outcomes; physical complaints, psychological functioning, family functioning and QoL. The data collection has been finalized in 2017.

ELIGIBILITY:
Inclusion Criteria:

* All participants in a family program

Exclusion Criteria:

* None

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Family members of patients in treatment for SUD at a Norwegian addiction treatment unit. The family members participated in a 4-day psychoeducational program
Sampling Method: Non-Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Caregiver burden | Changes from baseline to the 3 months follow-up
  Changes in Codependency symptomatology measured with the Composite Codependency Scale (CCS). Participants indicate the extent to which they agreed with each statement on a scale of 1 (strongly disagree) to 5 (strongly agree).
Family functioning | Changes from baseline to the 3 months follow-up
  Changes in the general family functioning subscale (GFFS). Respondents complete 12 items with a four-point response scale (1 = strongly agree, 4 = strongly disagree). A mean score is computed and a higher score indicated greater family dysfunction.

SECONDARY OUTCOMES:
Mental distress | Changes from baseline to the 3 months follow-up
  Changes in the the Hopkins Symptom Checklist (HSCL) 10-item version, which is used to measure mental distress. This 10-item index maps symptoms of anxiety (4 items) and depression (6 items) on 4-point Likert-type scales ranging from "not bothered at all" (1) to "extremely bothered" (4). The global severity index (GSI) constitutes the average of all items, with the highest score indicating greater symptom severity during the past week.
Physical complaints | Changes from baseline to the 3 months follow-up
  Changes in physical complaints, measured on a 10-point ordinal scale (scaled 0 - 10) with higher score indicating more complaints.
Well-being / quality of life | Changes from baseline to the 3 months follow-up
  Changes in Quality of Life measured with the QoL-5 scale (5 items). Responses are scored on a five-point scale ranging from very poor to very good QoL and then recoded into a decimal scale from 0.1 to 0.9, where 0.9 is the highest/best score and 0.1 the lowest/worst

CONTACTS AND LOCATIONS:
Overall Officials: John-Kåre Vederhus, PhD, Principal Investigator — Sørlandet Hospital
Locations (1):
- Addiction Unit - Sørlandet Hospital, Kristiansand, Agder, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vederhus JK, Kristensen O, Timko C. How do psychological characteristics of family members affected by substance use influence quality of life? Qual Life Res. 2019 Aug;28(8):2161-2170. doi: 10.1007/s11136-019-02169-x. Epub 2019 Mar 20. PMID 30895489